CLINICAL TRIAL: NCT01244009
Title: A Phase II Efficacy Study of MK-4827 in Patients With Mantle Cell Lymphoma
Brief Title: A Study of MK-4827 for the Treatment of Mantle Cell Lymphoma (MK-4827-002)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Tesaro, Inc. (Industry)
Responsible Party: Vice President of Late Stage Development, Merck Sharp & Dohme Corp
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MK-4827-002
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Last update posted 2016-11-07 (Estimated); Status verified 2016-11

CONDITIONS: Lymphoma; Mantle-Cell
Keywords: Poly (ADP-ribose) polymerase (PARP) inhibitor
MeSH Terms: conditions — Lymphoma | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MK-4827 (Experimental): All Participants
  Interventions: Drug: MK-4827

INTERVENTIONS:
Drug: MK-4827 — MK-4827 will be administered daily as an oral formulation in continuous 21-day cycles.

SUMMARY:
This study will investigate the efficacy and safety of MK-4827 in participants with relapsed mantle cell lymphoma (MCL) and in a subset of participants with inactivation of the Ataxia-Telangiectasia Mutated (ATM) gene.

ELIGIBILITY:
Inclusion Criteria :

* Participant must have a diagnosis of MCL that has relapsed after at least one prior chemotherapy regimen or for which the participant has refused standard therapy
* Participant has measureable disease defined by lymphadenopathy, organomegaly, bone marrow involvement and/or circulating lymphoma cells. At least one lesion must be > 2 cm in the longest diameter and measurable in 2 perpendicular dimensions
* Participant has a performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Female participants of child-bearing potential agree to use two approved contraceptive methods or remain abstinent throughout the study
* Male participants agree to use an adequate method of contraception throughout the study
* Participant has no history of prior cancer except certain cervical, skin, or prostate cancers, or has undergone potentially curative therapy with no recurrence for five years, or is deemed at low risk for recurrence
* Participant has not had any platelet or red blood cell transfusions or colony stimulating factor support during the month prior to treatment
* Participant has a pre-study diagnostic formalin fixed paraffin-embedded tumor tissue sample available

Exclusion Criteria :

* Participant has had chemotherapy, radiotherapy, or biological therapy within 4 weeks of screening
* Participant has a history of central nervous system (CNS) lymphoma
* Participant requires the use of corticosteroids
* Participant is pregnant, breastfeeding, or expecting to conceive or father children during the study
* Participant is known to be human immunodeficiency virus (HIV)-positive
* Participant has a history of Hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have a complete response (CR) or partial response (PR) during the study | Tumor assessments will be performed every 9 weeks for the first year the participant is on treatment, every 12 weeks in year 2, and every 6 months in year 3 and beyond

SECONDARY OUTCOMES:
Number of Participants with adverse events | From the day of enrollment through 30 days after the last dose of study drug
Time from allocation to disease progression or death from any cause (Progression-free survival) | Tumor assessments will be performed every 9 weeks for the first year the participant is on treatment, every 12 weeks in year 2, and every 6 months in year 3 and beyond